CLINICAL TRIAL: NCT02929030
Title: Safety and Efficacy of Polymer-free Sirolimus-eluting Coronary Stents in Patients With Coronary Artery Disease.
Brief Title: Clinical Performance of Nano Plus Sirolimus-Eluting Stents in Patients With Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Tao Ling, Professor, Xijing Hospital
Other Study IDs: NANOxijing001
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NANO Plus SES: All patients will be treated with NANO plus sirolimus-eluting stent. Patients will be prescribed with clopidogrel and aspirin before the index procedure. The lesions will be predilted if necessary before stent implantation. There are no specific limitations on coronary lesions according the study criteria.
  Interventions: Device: Nano

INTERVENTIONS:
Device: Nano — The stent system comprises of 2 components: stent steel platform, antiproliferative drug sirolimus, and stent balloon

SUMMARY:
The study aims to evaluate the safety and efficacy of polymer-free sirolimus-eluting coronary stent system (NANO plus) in patients with coronary artery disease . The primary endpoint is target lesion failure, a composite endpoint of cardiac death, target vessel related myocardial infarction and clinically-driven target lesion revascularization at 1 year follow-up.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single arm clinical registry investigating the safety and efficacy of polymer-free sirolimus-eluting coronary stent system (NANO plus) in patients with coronary artery disease . In total, we plan to recruit 2500 patients in real world setting. The patients will be followed clinically at 1-, 6- month and 1-, 2-, 3-, 4-, 5-year. All clinical data will be collected and managed by statistical center, clinical endpoint adjudication committee.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old, male or non-pregnancy female;
* Patients with coronary artery disease who match the indication of stent implantation;
* Patients who can understand the nature of the study, agree to participate and accept clinical follow-up;

Exclusion Criteria:

* Patients who can not tolerate the material or medication in this study;
* Pregnancy or lactation women
* Patients who had participated in another investigational drug or device trial that has not completed the primary endpoint;
* Patients are, in the opinion of the investigator, unable to comply with the requirements of the study protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
target lesion failure (TLF) | 12 months
  cardiac death, target vessel related myocardial infarction and/or clinically driven target lesion revascularization

SECONDARY OUTCOMES:
Target lesion failure | 1、6、12、24、36、48、60 months
  a composite endpoint of cardiac death, target lesion related myocardial infarction, and/or target lesion revascularization
Patient oriented composite endpoint | 1、6、12、24、36、48、60 months
  a composite endpoint of all cause death, all myocardial infarction and all revascularization
all cause death | 1、6、12、24、36、48、60 months
cardiac death | 1、6、12、24、36、48、60 months
Myocardial infarction | 1、6、12、24、36、48、60 months
Stent thrombosis | 1、6、12、24、36、48、60 months
Target lesion revascularization | 1、6、12、24、36、48、60 months
Target vessel revascularization | 1、6、12、24、36、48、60 months
target lesion failure | 1、6、24、36、48、60 months
  cardiac death, target vessel related myocardial infarction and/or clinically driven target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Lin Tao, PhD, Principal Investigator — Xijing Hospital; Yao-Jun Zhang, PhD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University; Yue Li, PhD, Principal Investigator — The First Clinical Hospital affiliated to Harbin Medical University; Zhiqi Sun, PhD, Principal Investigator — Daqing oilfield central hospital
Locations (1):
- Xijing Hospital, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Suwannasom P, Onuma Y, Benit E, Gach O, von Birgelen C, Hofma SH, Sotomi Y, Bo X, Zhang YJ, Gao R, Garcia-Garcia HM, Wykrzykowska JJ, de Winter RJ, Serruys PW. Evaluation of vascular healing of polymer-free sirolimus-eluting stents in native coronary artery stenosis: a serial follow-up at three and six months with optical coherence tomography imaging. EuroIntervention. 2016 Aug 5;12(5):e574-83. doi: 10.4244/EIJV12I5A97. PMID 27497357
- [Background] Zhang Y, Chen F, Muramatsu T, Xu B, Li Z, Ge J, He Q, Yang Z, Li S, Wang L, Wang H, He B, Li K, Qi G, Li T, Zeng H, Peng J, Jiang T, Zeng Q, Zhu J, Fu G, Bourantas CV, Serruys PW, Huo Y. Nine-month angiographic and two-year clinical follow-up of polymer-free sirolimus-eluting stent versus durable-polymer sirolimus-eluting stent for coronary artery disease: the Nano randomized trial. Chin Med J (Engl). 2014;127(11):2153-8. PMID 24890170
- [Derived] He X, Liu Y, Yin Z, Li F, van Geuns RJ, Garg S, Onuma Y, Serruys PW, Gao C, Tao L. Mid-term outcomes of paclitaxel-coated balloon for de novo non-small coronary lesions: a pooled analysis. BMC Med. 2025 Oct 31;23(1):598. doi: 10.1186/s12916-025-04429-9. PMID 41174582
- [Derived] Dai Y, Wang R, Chen F, Zhang Y, Liu Y, Huang H, Yang P, Zhang R, Zheng B, Gao C, Chen Y, Tao L. Clinical outcomes in 2481 unselected real-world patients treated with a polymer-free sirolimus-eluting stent: 3 years results from the NANO multicenter Registry. BMC Cardiovasc Disord. 2021 Nov 12;21(1):537. doi: 10.1186/s12872-021-02356-0. PMID 34772347
- [Derived] Liu Y, Zhang Y, Li Y, Qi T, Pan D, Wang H, Liu C, Ma D, Fang Z, Zhang R, Mou F, Tao L; NANO All-Comers Registry Investigators. One-year clinical results of the NANO registry: A multicenter, prospective all-comers registry study in patients receiving implantation of a polymer-free sirolimus-eluting stent. Catheter Cardiovasc Interv. 2020 Feb;95 Suppl 1:658-664. doi: 10.1002/ccd.28734. Epub 2020 Jan 21. PMID 31961057